CLINICAL TRIAL: NCT04329741
Title: Strengthening the Bond Between Owners and Their Dogs to Increase Physical Activity
Brief Title: The Stealth Pet Obedience Training Study
Acronym: SPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Grant #16-00293
Record Dates: First submitted 2019-10-04; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity
Keywords: dog walking; dog ownership; human-animal interaction
MeSH Terms: conditions — Motor Activity; Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 6-week basic dog obedience training course
  Interventions: Behavioral: 6-week basic dog obedience training course
- Control (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: 6-week basic dog obedience training course — The class focused on teaching owners how to better communicate with their dog and covered basic commands (e.g., sit, down, watch), loose leash walking, and polite greetings, among other skills. The importance of dog walking was implied, but not specifically emphasized. Classes were held once per week for 45 minutes, with 5-8 students per class.
  Arms: Intervention

SUMMARY:
Americans love pets. Nearly 1 in 2 American households (44%) own at least one pet dog and more than 1 in 3 (35%) own a cat. The bond people form with their pets can be powerful and can provide many mental and physical health benefits. In the case of pet dogs, a strong dog-owner bond increases the odds of regular dog walking, which can help owners meet physical activity guidelines. When the bond is strong, owners feel a sense of responsibility to walk the dog, as well as motivation and social support to walk. Dog walking may be a particularly sustainable form of physical activity as dogs require regular exercise throughout their lives, across all seasons. Owners less bonded to their dogs are less likely to walk them regularly and 40% of owners report never walking their dog.

Obedience training may strengthen the dog-owner bond. Thus, the proposed study will test the hypotheses that obedience training can 1) strengthen the dog-owner bond, and 2) promote physical activity among owners. Forty dog owners who do not regularly walk their dog will be randomized to a 6-week obedience training course (n=20) or a control group that does not receive dog training (n=20). The investigators will assess the strength of the dog-owner bond (via questionnaires) and physical activity levels (via a wearable activity monitor) before training, immediately after completing training, and 6 weeks after completing training. The hypothesis is that the dog-owner bond will strengthen and physical activity levels will increase in the intervention group as compared to the control group. As over 50 million American households own a dog, support for this hypothesis would support further investigation of dog obedience training as a novel strategy for promoting public health.

ELIGIBILITY:
Inclusion Criteria:

* Age 21+ years
* Current dog owner
* Walk dog ≤3 for no more than 20 minutes
* Have not attended obedience training course
* English speaking

Exclusion Criteria:

* Have a dog with a history of aggressive behavior
* Have a dog overdue for rabies vaccination (self-reported)
* Self-report regular exercise over last 6 months
* Have any condition that limits walking ability
* Have uncontrolled hypertension or diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in physical activity from baseline to 6 weeks | 7 days at baseline, 6 weeks
  Measured with ActiGraph wGT3X-BT accelerometers
Change in physical activity from baseline to 12 weeks | 7 days at baseline, 12 weeks
  Measured with ActiGraph wGT3X-BT accelerometers

SECONDARY OUTCOMES:
Change in sedentary behavior from baseline to 6 weeks | 7 days at baseline, 6 weeks
  Measured with ActiGraph wGT3X-BT accelerometers
Change in sedentary behavior from baseline to 12 weeks | 7 days at baseline, 12 weeks
  Measured with ActiGraph wGT3X-BT accelerometers
Change in dog-owner bond strength from baseline to 6 weeks | baseline, 6 weeks
  The Perceived Emotional Closeness sub-scale of the Cat/Dog Owner Relationship Scale (C/DORS) was used to assess dog-owner bond strength. The sub-scale score can range from 1-5, with a higher score indicating greater emotional closeness.
Change in dog-owner bond strength from baseline to 12 weeks | baseline, 12 weeks
  The Perceived Emotional Closeness sub-scale of the Cat/Dog Owner Relationship Scale (C/DORS) was used to assess dog-owner bond strength. The sub-scale score can range from 1-5, with a higher score indicating greater emotional closeness.
Change in dog walking self-efficacy from baseline to 6 weeks | baseline, 6 weeks
  Sub-scales from the Dogs and Walking Survey (DAWGS) were used to assess social cognitive theory-based determinants of dog walking behavior. The self-efficacy sub-scale is scored on a scale of 9-45, with higher scores indicating greater dog walking self-efficacy.
Change in dog walking self-efficacy from baseline to 12 weeks | baseline, 12 weeks
  Sub-scales from the Dogs and Walking Survey (DAWGS) were used to assess social cognitive theory-based determinants of dog walking behavior. The self-efficacy sub-scale is scored on a scale of 9-45, with higher scores indicating greater dog walking self-efficacy.
Change in social support for dog walking from baseline to 6 weeks | baseline, 6 weeks
  Sub-scales from the Dogs and Walking Survey (DAWGS) were used to assess social cognitive theory-based determinants of dog walking behavior. The social support for dog walking sub-scale is scored on a scale of 3-15, with higher scores indicating greater perceived support from one's dog for walking.
Change in social support for dog walking from baseline to 12 weeks | baseline, 12 weeks
  Sub-scales from the Dogs and Walking Survey (DAWGS) were used to assess social cognitive theory-based determinants of dog walking behavior. The social support for dog walking sub-scale is scored on a scale of 3-15, with higher scores indicating greater perceived support from one's dog for walking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No